CLINICAL TRIAL: NCT01647321
Title: Evaluating the Effects of Functional Electrical Stimulation on Ambulation in Individuals With Secondary Progressive Multiple Sclerosis
Brief Title: Functional Electrical Stimulation for Individuals With Secondary Progressive Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NA_00069253
Record Dates: First submitted 2012-07-19; First posted 2012-07-23 (Estimated); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Secondary Progressive Multiple Sclerosis
Keywords: SPMS
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive | interventions — Endurance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active cycling (Active Comparator): Individuals will receive functional electrical stimulation while on the stationary bike and instructed to actively pedal.
  Interventions: Behavioral: Active cycling
- Passive cycling (Sham Comparator): Individuals will receive active functional electrical stimulation (FES) while on the stationary bike and instructed to relax their legs, allowing the FES to move their legs on the stationary bike.
  Interventions: Behavioral: Passive cycling

INTERVENTIONS:
Behavioral: Active cycling — The exercise program uses a stationary bike equipped with functional electrical stimulation (FES) of leg muscles. Participants are instructed to actively pedal while the FES is assisting. The training program is expected to be performed for one hour, three times a week for 12 weeks.
  Other Names: cycling; endurance training
  Arms: Active cycling
Behavioral: Passive cycling — The exercise program uses a stationary bike equipped with functional electrical stimulation (FES) of leg muscles. Participants are instructed to sit passively on the stationary bile while the FES is assisting. The training program is expected to be performed for one hour, three times a week for 12 weeks.
  Other Names: letting the functional electrical stimulation move the legs
  Arms: Passive cycling

SUMMARY:
Secondary progressive multiple sclerosis (SPMS) is a subtype of multiple sclerosis (MS) for which there are no existing therapies that alter the disease course. This research will utilize cutting edge functional electrical stimulation (FES) cycling technology with the goal of improving walking in individuals with SPMS. The investigators hypothesize that FES cycling will improve walking in subjects with SPMS.

DETAILED DESCRIPTION:
Individuals with secondary progressive multiple sclerosis (SPMS) experience significant impairments in ambulation leading to use of canes, walkers, and ultimately wheelchairs. Treatment attempts for progressive MS have been disappointing. No therapeutic intervention has been shown to modulate disability in patients with SPMS. FES cycling has been shown to have multiple primary medical benefits including: increased muscle mass, improvements in bone density, enhanced cardiovascular function, improved bowel function, decreased spasticity and reductions in bladder infection rate. More importantly FES may modulate the inflammatory central nervous system (CNS) environment in progressive MS. The investigators are proposing a novel, and easy to implement intervention strategy of FES cycling to help improve gait function in individuals with SPMS. A successful outcome on a larger SPMS population would have significant impact towards changing MS clinical care. FES is easily transferable to clinical practice and could potentially ameliorate other complications associated with SPMS such as spasticity, mood and fatigue reducing the burden of health care cost. In addition, the investigators will gain a better understanding of the mechanisms underlying these changes that could be used to design new therapeutic strategies.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of secondary progressive multiple sclerosis
* males and females between the ages of 18 and 65 years
* Expanded disability status scale score between 5.0 and 7.0
* Able to consent to participate in study and are willing to undergo a lumbar puncture and blood draws
* If on on Ampyra or anti-spasticity agent, must be on stable dose for 1 month prior to screening
* No functional electrical stimulation use within 4 weeks
* Participants must be medically stable with no recent (1 month or less) inpatient admission for acute medical or surgical issues

Exclusion Criteria:

* Uncontrolled hypertension or other significant cardiovascular disease as determined by investigator
* History of epileptic seizures
* Subjects who have a pacemaker
* Relapse within thirty days prior to screening visit
* Pregnancy
* Subjects having a Stage 2 or greater sacral decubitus ulcer

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Change in timed 25 foot walk from baseline to end of training | Participants are assessed at baseline (visit 1), one-month (visit 2), two-months (visit 3), three-months (visit 4), end of study (visit 5)
  Here we will assess whether a subjects walking speed is improved following active cycling with functional electrical stimulation. Our prediction is that individuals will improve in their walking function following seated active cycling with functional electrical stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Newsome, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins / Kennedy Krieger Institute, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No